Last update: 01/02/2018

Development of a National, Evidence Based Protocol for Stroke Rehabilitation in a Multicenter Italian no Profit Institution: Implementation and Results of a Pilot Study

## Statistical analysis

Data were analysed using IBM SPSS Statistics 24.0 for Windows. Shapiro-Wilk test was used to verify if parameters were normally distributed (significance level set to 5%). According to the test results, parameters characterized by a normal distribution were represented by mean and standard deviation, parameters with a non-normal distribution by median and interquartile range, dichotomous parameters by percentage. Clinical and functional parameters measured at admission were compared to those measured at discharge by using a paired t-test for continuous, normally distributed variables, a Wilcoxon signed rank test for ordinal and not normally distributed variables and a McNemar test for dichotomous variables. A p-value < 0.05 was chosen for statistical significance.